CLINICAL TRIAL: NCT00025987
Title: Thermal Responses In Normal Volunteers To Head-Neck Cooling
Brief Title: Temperature Response to a Head-Neck Cooling System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020025; 02-N-0025
Record Dates: First submitted 2001-11-02; First posted 2001-11-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Healthy
Keywords: Brain; Temperature; Lower; Tympanic; Rectal; Cooling of the Head and Neck; Control; Epilepsy; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy | interventions — Thermometers

INTERVENTIONS:
Device: Head and Neck Cooling System
Device: Thermometer Pill

SUMMARY:
This study will evaluate the effectiveness of a specially designed head-neck cooling system for way lowering the body's central, or core, temperature and cooling the brain. Brain cooling has an effect on stopping seizure discharges in the brain as well as the seizures themselves. If this system works to cool the brain, a similar study may be tried in patients with epilepsy.

Normal volunteers 21 years of age and older who have no medical or neurological condition and do not use any medications may be eligible for this study. Candidates will be screened with an interview. Women will have a pregnancy test. Those enrolled will be hospitalized twice for overnight stays, with the admissions 2 to 3 days apart.

Participants will have a medical history, physical and neurological examinations, electroencephalogram (EEG) and electrocardiogram (EKG). Then, electrodes will be attached to their scalp, forearm and calf to measure temperatures in those locations. Intestinal (core) temperature will be measured with a temperature-sensing pill, which will be swallowed earlier), and a hand-held infrared thermometer will be used to measure temperatures from the ear canal, face, head, arms legs, and abdomen. Electrodes on the scalp will also measure changes in blood volume in the brain for a study of brain blood flow. Subjects will be seated in a comfortable chair and fitted with the cooling system, a portable unit with a circulating coolant. Cooling will last 30 minutes for the first session and 60 minutes for the second. Participants will be monitored for at least 30 minutes after each session to track temperature changes and have a post-cooling EEG recording.

DETAILED DESCRIPTION:
The aim of this protocol is to study thermal responses in normal volunteers using a special cooling system designed to cool the head and neck. Temperature will be monitored at various locations including the scalp, face, mouth, ears (tympanic), arms, legs, and rectum. Previous studies indicate that cooling of the brain can be achieved with the head-neck cooling method. We hope to derive cooling parameters that will be used in a future study involving patients with epilepsy.

ELIGIBILITY:
INCLUSION CRITERIA:

21 years and older

No neurological or medical condition

No use medication of any kind, including prescription, over-the-counter or herbal medicines.

No history of any kind of gastrointestinal tract disorders

EXCLUSION CRITERIA:

Women who are pregnant (screened with urine pregnancy test)

Those with progressive neurological disorders

Those sensitive to coldness

Those taking medication

Those who smoke

Those whose heart rate less than 50 or more than 100

Those who are less than 80 pounds or excessively overweight

Those who have a history of gastrointestinal disorders (i.e. diverticulitis and other inflammatory bowel diseases)

Those who have difficulty swallowing or whose gag reflex is impaired

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2001-11; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Amoateng-Adjepong Y, Del Mundo J, Manthous CA. Accuracy of an infrared tympanic thermometer. Chest. 1999 Apr;115(4):1002-5. doi: 10.1378/chest.115.4.1002. PMID 10208200
- [Background] Ao H, Moon JK, Tanimoto H, Sakanashi Y, Terasaki H. Jugular vein temperature reflects brain temperature during hypothermia. Resuscitation. 2000 Jul;45(2):111-8. doi: 10.1016/s0300-9572(00)00154-4. PMID 10950319
- [Background] Baumgartner FJ, Janusz MT, Jamieson WR, Winkler T, Burr LH, Vestrup JA. Cardiopulmonary bypass for resuscitation of patients with accidental hypothermia and cardiac arrest. Can J Surg. 1992 Apr;35(2):184-7. PMID 1562930